CLINICAL TRIAL: NCT06747663
Title: Reliability of MRI and Ultrasound in Predicting Needle Depth During Cervical Epidural Injections: a Methodological Observational Study
Brief Title: Reliability of MRI and Ultrasound in Cervical Epidural Needle Depth Estimation
Acronym: CERV-MRI-USG
Status: Not yet recruiting | Type: Observational
Sponsor: Damla Yürük (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Damla Yürük, Associate Professor of Algology, Diskapi Teaching and Research Hospital
Organization: Diskapi Teaching and Research Hospital (Other)
Other Study IDs: Ankara Etlik City Hospital; AEŞH-BADEK-2024-1133 (Registry Identifier: Ankara City Hospital Ethics Committee AEŞH-BADEK-2024-1133 Approval Date: 27.11.2024)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Neck Pain; Radicular Pain; Cervical Epidural Injection
Keywords: Cervical Epidural Steroid Injection; Needle Depth Estimation; Ultrasound Guidance; MRI Guidance; Fluoroscopy; Radiation Exposure; Chronic Pain Management
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cervical Epidural Injection Group: Participants undergoing cervical epidural injections for chronic neck and radicular pain. Needle depth will be measured pre-procedurally using MRI and ultrasound and compared with fluoroscopy-guided needle placement to assess reliability and radiation exposure.
  Interventions: Procedure: Needle Depth Measurement Using MRI, Ultrasound, and Fluoroscopy

INTERVENTIONS:
Procedure: Needle Depth Measurement Using MRI, Ultrasound, and Fluoroscopy — This intervention involves cervical epidural steroid injection (CESI) for patients with chronic neck and radicular pain. Needle depth is measured pre-procedurally using MRI and ultrasound to predict the ideal needle placement. Fluoroscopy is used during the procedure to confirm and compare these measurements, aiming to evaluate the accuracy of imaging techniques and minimize radiation exposure.

SUMMARY:
This study aims to evaluate the reliability of magnetic resonance imaging (MRI) and ultrasound (USG) in predicting needle depth during cervical epidural injections, compared to fluoroscopy. The goal is to identify alternative imaging methods that reduce radiation exposure while maintaining procedural accuracy and patient safety.

DETAILED DESCRIPTION:
Cervical epidural steroid injections (CESI) are commonly used to manage chronic neck and radicular pain. Accurate needle placement is critical for the success and safety of the procedure. Fluoroscopy is the standard method for guiding the needle; however, it exposes patients and clinicians to ionizing radiation.

This study compares pre-procedural MRI and USG measurements of needle depth with fluoroscopy-guided needle depth during CESI.

Primary Objective: Assess the agreement between MRI, USG, and fluoroscopy measurements of needle depth using intraclass correlation coefficients (ICC) within a ±0.3 cm tolerance.

Secondary Objectives: Evaluate the correlation between fluoroscopic lateral imaging frequency and radiation exposure.

The study is a methodological observational study conducted at Ankara Etlik City Hospital, involving adult patients undergoing CESI. Data will be collected retrospectively and prospectively for eligible participants.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years, Diagnosed with chronic cervical pain, Referred for cervical epidural steroid injection, Patients capable of providing informed consent.

Exclusion Criteria:

Age < 18 years, Pregnancy or breastfeeding, History of coagulation disorders or use of anticoagulants, Severe systemic infections or local infections at the injection site, Known allergy to steroids or local anesthetics, Uncontrolled diabetes mellitus, Patients with spinal tumors or significant spinal deformities, Previous cervical spine surgery, Cognitive impairment preventing informed consent or follow-up participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 years and older, diagnosed with chronic cervical pain, and referred for cervical epidural steroid injection. Patients must be capable of providing informed consent and participating in follow-up assessments. Individuals with contraindications such as pregnancy, severe systemic infections, coagulopathy, known allergies to steroids or anesthetics, or prior cervical spine surgery are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Needle Depth Prediction Using MRI and Ultrasound Compared to Fluoroscopy in Cervical Epidural Steroid Injections | 1 day (during the procedure)
  The primary outcome measure evaluates the reliability and accuracy of pre-procedural needle depth measurements obtained using MRI and ultrasound imaging compared to intra-procedural fluoroscopy during cervical epidural steroid injections. The goal is to determine the concordance between these imaging techniques and assess their utility in reducing procedural radiation exposure.

SECONDARY OUTCOMES:
Radiation Exposure During Cervical Epidural Steroid Injections | 1 day (during the procedure)
  The secondary outcome measure assesses the level of radiation exposure (in mGy) experienced by patients and practitioners during cervical epidural steroid injections when fluoroscopy is used. Comparisons will be made to determine if the use of pre-procedural MRI or ultrasound reduces fluoroscopy duration and radiation exposure.

CONTACTS AND LOCATIONS:
Overall Officials: DAMLA YÜRÜK, Associate Professor of Algolog, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to concerns regarding patient confidentiality and data privacy regulations. Data sharing is not part of the current study plan

REFERENCES:
- [Background] Pak MH, Lee WH, Ko YK, So SY, Kim HJ. Ultrasonographic measurement of the ligamentum flavum depth; is it a reliable method to distinguish true and false loss of resistance? Korean J Pain. 2012 Apr;25(2):99-104. doi: 10.3344/kjp.2012.25.2.99. Epub 2012 Apr 4. PMID 22514777